CLINICAL TRIAL: NCT05162963
Title: Impact of Implant-supported Removable Prosthesis Versus Fixed Prosthesis on Quality of Life in Edentulous Patients: a Multicenter Non-inferiority Cross-over Trial
Brief Title: Impact of Removable Versus Fixed Implant-supported Prostheses in Oral Health Quality of Life for Edentulous Patients
Acronym: FALBALA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: APHP210087
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-05

CONDITIONS: Complete Edentulism
Keywords: Overdenture; Complete edentulism; Quality of life; Dental implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with fixed implant denture (Active Comparator): Patients quality of life will be compared when using a removable implant denture and a fixed implant denture, in a cross-over design. Fixed denture is considered the standard protocol.
  Interventions: Other: fixed implant denture; Other: removable implant denture
- Patients treated with removable implant denture (Experimental): Patients quality of life will be compared when using a removable implant denture and a fixed implant denture, in a cross-over design. Removable denture is considered the experimental protocol.
  Interventions: Other: fixed implant denture; Other: removable implant denture

INTERVENTIONS:
Other: fixed implant denture — Patients will receive four or six dental implants, four in the mandible or six in the maxilla, depending on the arch to be treated. After an osseointegration phase of 4 to 6 months, two implant prostheses will be made for each patient, one removable, the other fixed. According to the randomization, during an initial period of 6 months, half of the patients will be using the removable prosthesis, the other half the fixed prosthesis. A 15-day washout will be performed. Then, during a second period of 6 months, the patients will be using the second prosthesis.
Other: removable implant denture — removable implant denture

SUMMARY:
Comparison between fixed and removable implant-retained complete prostheses previously showed that while patients appreciate the ergonomic cleaning of removable prostheses, they prefer the comfort and masticatory efficiency of fixed prostheses. New treatment strategies are emerging; the use of telescopic attachments now offers a prosthetic alternative for the treatment of edentulous teeth at a lower financial cost than fixed prostheses.

To answer this question, the study is constructed as a cross-over. 30 patients will use a removable telescopic prosthesis and then a fixed prosthesis, or vice versa, for a period of 6 months according to randomization. They will answer a quality of life questionnaire after each period and finally choose their favorite prosthesis. The null hypothesis is that removable telescopic implant prostheses will result in a quality of life comparable to that obtained with fixed implant-supported prostheses.

The primary objective of this study is to demonstrate the non-inferiority of removable versus fixed prostheses on quality of life after 6 months of use of each implant-supported prosthesis in edentulous maxillary or mandibular patients. The measurement of the evolution of the quality of life is analyzed using the GOHAI questionnaire after 6 months of use of each prosthesis.

The secondary objectives are to:

* Determine the decisional parameters in the final choice of the prosthesis by the patient at the end of the study, with the Mc Gill Denture Satisfaction Instrument,
* Compare the masticatory efficiency between the two dentures (duration, number of cycles and frequency of chewing of the carrot test food, with each denture after 6 months of use),
* Compare the oral hygiene between the two prostheses (peri-implant plaque index, after 6 months for each prosthesis),
* Compare the adjustments and repair required after the placement of each prosthesis and the chairside treatment time to achieve them,
* Compare the complications and their frequency of occurrence with each type of prosthesis during the 6-month wearing period.

DETAILED DESCRIPTION:
Edentulism is defined as the loss of all natural teeth and is an important public health issue globally for its high prevalence (exceeding 10% in adults aged ≥ 50 years) and associated disability Epidemiological studies show a decrease in the prevalence of total edentulism but an increase in the number of edentulous people in the world in general and in Western society in particular, linked to the increase in life expectancy. In Europe, the edentulism rate varies greatly from one country to another. According to the WHO, in the 65+ age group, the rate of total edentulism in 2000 was 60-70% in some European countries and still 15% in France.

Prosthetic rehabilitation is a factor of social inequalities in health insofar as this care is poorly covered or not covered by social organizations. The different treatment solutions must be examined in terms of the gain they represent in terms of quality of life compared to their cost.

The improvement of retention of a removable prosthesis with implants was demonstrated. The comparison between fixed and removable implant-retained prostheses previously showed that while patients appreciate the ergonomic cleaning of removable prostheses, they prefer the comfort and masticatory efficiency of fixed prostheses. New treatment strategies are emerging; the use of telescopic attachments now offers a prosthetic alternative for the treatment of edentulous teeth at a lower financial cost than fixed prostheses. This treatment option is not well known. There are no randomized controlled studies directly comparing these two therapies in terms of quality of life.

To answer this question, the study is constructed as a cross-over. 30 patients will use a removable telescopic prosthesis and then a fixed prosthesis, or vice versa, for a period of 6 months according to randomization. They will answer a quality of life questionnaire after each period and finally choose their favorite prosthesis. The null hypothesis is that removable telescopic implant prostheses will result in a quality of life comparable to that obtained with fixed implant-supported prostheses.

The primary objective of this study is to demonstrate the non-inferiority of removable versus fixed prostheses on quality of life after 6 months of use of each implant-supported prosthesis in edentulous maxillary or mandibular patients. The measurement of the evolution of the quality of life is analyzed using the GOHAI questionnaire after 6 months of use of each prosthesis, i.e. twice during the study.

The GOHAI is a specific oral quality of life scale, comprising 12 items scored from 1 to 5 divided into 3 subparts corresponding to the functions of speaking, eating, and swallowing, psychosocial aspects, and pain/discomfort. A score of 60 corresponds to an optimal quality of life.

The secondary objectives are to:

* Determine the decisional parameters in the final choice of the prosthesis by the patient at the end of the study, with the Mc Gill Denture Satisfaction Instrument,
* Compare the masticatory efficiency between the two dentures (duration, number of cycles and frequency of chewing of the carrot test food, with each denture after 6 months of use),
* Compare the oral hygiene between the two prostheses (peri-implant plaque index, after 6 months for each prosthesis),
* Compare the adjustments and repair required after the placement of each prosthesis and the chairside treatment time to achieve them,
* Compare the complications and their frequency of occurrence with each type of prosthesis during the 6-month wearing period.

Experimental design All patients will receive four or six dental implants, four in the mandible or six in the maxilla, depending on the arch to be treated. After an osseointegration phase of 4 to 6 months, two implant prostheses will be made for each patient, one removable, the other fixed. All patients will receive specific training in oral and peri-implant hygiene. According to the randomization, during an initial period of 6 months, half of the patients will be using the removable prosthesis, the other half the fixed prosthesis. A 15-day washout will be performed. No residual effect are expected, but the assessment of the baseline quality of life require daily use of the conventional prosthesis (without implant). Then, during a second period of 6 months, the patients will be using the second prosthesis. At the end of the study, the patient will choose the prosthesis he prefers and justifies his choice in a specific questionnaire.

A measurement of quality of life (GOHAI questionnaire) will be carried out before treatment and after use of each type of prosthesis. At the 6-month appointment of each prosthesis, evaluations will be performed including a plaque index measurement and a masticatory efficiency test. The adjustments and repairs required during the time the prosthesis will be worn, as well as the time required to perform them, will be recorded. A follow-up of the complications that occurred on each type of prosthesis will be set up during the two prosthetic phases.

The analysis will be carried out in intention-to-treat and per-protocol analysis. The treatment effect will be estimated by the difference in the evolution of the GOHAI score between the period with a removable prosthesis and the period without a removable prosthesis and its 95% confidence interval. A sequence and carry over effect will be sought.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age;
* Mandibular AND/OR maxillary edentulous patients, treated with satisfying conventional denture for a minimum of 3 months;
* Bone volume compatible with the placement of implants of at least 9 mm in length;
* Sufficient inter-arch space;
* Free and informed consent;
* Affiliated to the social security fund.

Exclusion Criteria:

* Systemic pathologies contraindicating the placement of implants (unbalanced diabetes, biphosphonates);
* Smoking patient > 10 cigarettes per day;
* Class IV bone according to the Leckholm and Zarb classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the evolution of the quality of life using the GOHAI questionnaire | 6 months
  Measurement of the evolution of the quality of life is analyzed using the GOHAI questionnaire

SECONDARY OUTCOMES:
Scores of the Mc Gill Denture Satisfaction Instrument | 21 months
  Scores of the Mc Gill Denture Satisfaction Instrument, for the final choice of prosthesis, at the end of the study.
Measurement of the duration of chewing of the carrot test food | 6 months
  Measurement of the duration of chewing of the carrot test food at the swallowing threshold, after 6 months, for each prosthesis;
Measurement of the number of cycles of chewing of the carrot test food | 6 months
  Measurement of the number of cycles and frequency of chewing of the carrot test food at the swallowing threshold, after 6 months, for each prosthesis;
Measurement of the frequency of chewing of the carrot test food | 6 months
  Measurement of the frequency of chewing of the carrot test food at the swallowing threshold, after 6 months, for each prosthesis;
Peri-implant plaque index | 6 months
  Peri-implant plaque index (measured by the Mombelli score), after 6 months for each prosthesis
Adjustments required after placement | 6 months
  Adjustments required after placement, with each prosthesis (subprosthetic injuries, premature and occlusal interferences, retouching of the prosthetic intrados or extrados, adjustment of the retention force, modification of the prosthetic profile), during the 6-month wearing period for each prosthesis; The time of adjustment is measured from the moment the patient sits in the dental chair to the moment he/she leaves the chair, the unit is the quarter hour;
Complications | 6 months
  Complications (screw fractures, prosthetic screw loosening, ceramic fracture, prosthetic base fracture, attachment loss, abutment screw loosening, implant loss), during the 6-month wearing period, for each prosthesis.

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION